CLINICAL TRIAL: NCT01032408
Title: A Phase 3, Randomized, Controlled, Open Label Study to Evaluate the Immunogenicity, Safety, and Tolerability of MF59-Adjuvanted Versus Non-Adjuvanted Vaccines Against Novel H1N1 Virus in Patients With Human Immunodeficiency Virus Type 1 (HIV-1) Infection
Brief Title: Immunogenicity, Safety, and Tolerability of MF59-Adjuvanted Versus Non-Adjuvanted Influenza Vaccines in Patients With HIV-1 Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiltern Pesquisa Clinica Ltda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V111_14TP
Record Dates: First submitted 2009-12-14; First posted 2009-12-15 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: H1N1 Influenza Virus; Human Immunodeficiency Virus Type 1 (HIV-1) Infection
Keywords: Influenza A Virus; Virus Diseases; Influenza, Human; HIV-1; Immunodeficiency Virus; H1N1; HIV Infection; Immunogenicity; safety; tolerability
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections; Virus Diseases; Influenza, Human; HIV Infections | interventions — focetria

ARMS (4):
- HIV-1 Infected Subjects Receiving Vaccine with Adjuvant (Experimental): Each subject received two doses of vaccine with adjuvant (Focetria®), the first on Study Day 1, and the second on Study Day 22
  Interventions: Biological: Focetria®
- HIV-1 Infected Subjects Receiving Vaccine without Adjuvant (Experimental): Each subject received two doses of vaccine without adjuvant (Begrivac®), the first on Study Day 1, and the second on Study Day 22
  Interventions: Biological: Begrivac®
- Healthy Subjects Receiving Vaccine with Adjuvant (Experimental): Each subject received two doses of vaccine with adjuvant (Focetria®), the first on Study Day 1, and the second on Study Day 22
  Interventions: Biological: Focetria®
- Healthy Subjects Receiving Vaccine without Adjuvant (Experimental): Each subject received two doses of vaccine without adjuvant (Begrivac®), the first on Study Day 1, and the second on Study Day 22
  Interventions: Biological: Begrivac®

INTERVENTIONS:
Biological: Focetria® — 7.5 ug of HA antigen; adjuvanted; monovalent
  Arms: HIV-1 Infected Subjects Receiving Vaccine with Adjuvant; Healthy Subjects Receiving Vaccine with Adjuvant
Biological: Begrivac® — 15 ug of HA antigen; non-adjuvanted; trivalent
  Arms: HIV-1 Infected Subjects Receiving Vaccine without Adjuvant; Healthy Subjects Receiving Vaccine without Adjuvant

SUMMARY:
This is a phase III, randomized, controlled, open label study with two vaccine regimens. The study will assess the relative safety and immunogenicity of vaccine regimens comparing adjuvanted versus non-adjuvanted formulations of A(H1N1) inactivated influenza virus vaccine in subjects with Human Immunodeficiency Virus Type 1 (HIV-1) Infection and to compare safety and immunogenicity data with a contemporaneously enrolled control group of age-comparable, healthy subjects.

Because certain individuals may be hypo-responsive to influenza vaccination, additional studies with high-risk groups are warranted in order to determine the optimal vaccine formulation and dosing schedule for prevention of novel H1N1 virus infection.

ELIGIBILITY:
Inclusion Criteria:

For HIV-1 Infected Subjects:

* Adults between 18-60 years old (inclusive)
* Any sex or ethnicity
* Confirmed Diagnosis of HIV-1 infection
* CD4+ cells count >200 per mm3 within 3 months prior to inclusion in the study
* HIV-1 viral load below 200 copies/mL within 90 days prior to inclusion in the study
* Childbearing potential women must be willing to use an acceptable contraceptive method. Acceptable contraceptive methods are defined as one or more of the following:

  1. Hormone contraceptive (such as oral, injectable, transdermal patch, subcutaneous implant, cervical ring)
  2. Barrier (condom with spermicide or diaphragm with spermicide) at each intercourse and during the whole intercourse
  3. Intra-uterine device (IUD)
  4. Monogamous relation with vasectomized partner (must have been vasectomized at least six months before the volunteer entered the study)
* No changes in the antiviral therapy (including HAART) for the previous 4 weeks and/or change in the predicted antiviral therapy through study Day 43 (3 weeks after the second dose of the vaccine)
* No use of immunomodulatory therapy, including cyclosporine, interleukins, interferons, or systemic glucocorticoids (including inhalatory) within 3 months before study inclusion
* Subjects capable of respecting all the study procedures and available for all visits scheduled to the investigation site
* Subjects capable of understanding the nature and risk of the study proposed and signing the consent form
* The subjects may have other underlying diseases, such as, but not limited to, hypertension, diabetes, cardiac ischemic disease, or hypothyroidism, however their symptoms/signs must be currently under control with medical treatment according to the investigator's evaluation

For Healthy Adults:

* Adults between 18-60 years old (inclusive)
* Any sex and ethnicity
* Subjects with good health as determined by medical history, physical evaluation, and investigator's clinical opinion
* Childbearing potential women must be willing to use an acceptable contraceptive method. Acceptable contraceptive methods are defined as one or more of the following:

  1. Hormone contraceptive (such as oral, injectable, transdermal patch, subcutaneous implant, cervical ring).
  2. Barrier (condom with spermicide or diaphragm with spermicide) at each intercourse and during the whole sexual intercourse
  3. Intra-uterine device (IUD)
  4. Monogamous relation with vasectomized partner (must have been vasectomized for at least six months before the volunteer entered the study)
* Subjects capable of respecting all the study procedures and available for all the visits scheduled at the investigation site
* Subjects capable of understanding the nature and risk of the study proposed and signing the consent form

There will be NO blood sample collection of healthy volunteers viewing the determination of their serological status regarding the HIV virus.

Exclusion Criteria:

For HIV-1-Infected Subjects:

* HIV-1 viral load above 500 copies/mL within 6 months prior to inclusion in the study
* Previous laboratory confirmed diagnosis of an infection by the novel H1N1 virus
* Receipt of another vaccine against the novel H1N1 virus within 3 months prior to inclusion in the study
* Any recent vaccine given within the last 21 days (inclusive)
* History of allergic reaction to an influenza vaccine in the past, or a current or previous occurrence of allergy to egg or egg protein, kanamycin, and neomycin sulfate
* Acute febrile disease (vaccination may be delayed up to 3 days after the resolution of the symptoms)
* History of cancer, except for skin cancer, including Kaposi's Sarcoma, basal cell carcinoma, and non-invasive malignancy related to HPV
* History of cognitive disorders
* History of progressive or severe neurological disorders, including Guillain-Barré Syndrome
* Pregnancy or breast-feeding
* Use of immunomodulatory therapy, including cyclosporin, interleukins, and interferons, within 3 months prior to inclusion in the study
* Receipt of parenteral immunoglobulin, hemotherapy, and/or plasma derivatives within 3 months prior to inclusion in the study
* Projected life expectancy lower than 12 months
* Receipt of any investigational product within 12 months prior to inclusion in the study

For Healthy Adults:

* Previous laboratory confirmed diagnosis of an infection by the novel H1N1 virus
* Receipt of another vaccine against the novel H1N1 virus within 3 months prior to inclusion in the study
* Any recent vaccine given within the last 21 days (inclusive)
* History of allergic reaction to influenza vaccine in the past, or a current or previous allergy to egg or egg protein, kanamycin, and neomycin sulfate
* Acute febrile disease (the vaccination may be delayed up to 3 days after symptoms resolution)
* Pregnancy or breast-feeding
* Receipt of parenteral immunoglobulin, hemotherapy, and/or plasma derivatives within 3 months prior to inclusion in the study
* Receipt of any investigational product within 12 months prior to inclusion in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 154 (Actual)
Dates: Start 2010-04; Primary Completion 2011-09 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Geometric Mean HI Titer by Visit | 13 months after vaccination (Day 1, Day 22, Day 43, Day 133, Day 223 and Day 403)
  Geometric mean hemagglutination inhibition (HI) titer = GMT
Percentage of Subjects Who Reached Seroprotection by Visit | 13 Months after vaccination (Day 22, Day 43, Day 133, Day 223 and Day 403)
  The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with HIV infection.
  The percentage of subjects that reached seroprotection in comparison to the pre-vaccination result are presented by visit. Seroprotection was defined as HI titer ≥40.
Difference in the Seroconversion Rates or Significant Increase by Visit (Vaccine With Adjuvant - Vaccine Without Adjuvant) | 13 Months after vaccination (Day 22, Day 43, Day 133, Day 223 and Day 403)
  The primary objective of this study was to help determine the ideal strategy of vaccination against pandemic H1N1 influenza in subjects with invasive solid tumors/hematologic neoplasms.
  Comparisons were made by vaccine group using differences in the percentage of subjects with seroconversion/significant increase and were presented with 95% confidence intervals.

SECONDARY OUTCOMES:
Geometric Mean Ratio by Visit | 13 months after vaccination (Day 22/Day1, Day 43/Day 1, Day 43/Day 22, Day 133/Day 43, Day 223/Day 43 and Day 403/Day 223)
  The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with HIV infection.
Ratio of Immunogenicity Data by Visit (Vaccine with Adjuvant:Vaccine Without Adjuvant) | 13 months after vaccination (Day 1, Day 22, Day 22/Day1, Day 43, Day 43/Day 1, Day 43/Day 22, Day 133, Day 133/Day 43, Day 223, Day 223/Day 43 and Day 403, Day 403/Day 223)
  The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with HIV infection. Comparisons were made by vaccine group using ratios of immunogenicity data and were presented with 95% confidence intervals.
Percentage of Subjects Who Seroconverted or Had a Significant Increase in GMT by Visit | 13 Months after vaccination (Day 22, Day 43, Day 133, Day 223 and Day 403)
  The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with HIV infection.
  The percentage of subjects that reached seroconversion or had a significant increase in comparison to the pre-vaccination result were presented by visit. Seroconversion or a significant increase was defined as HI titer ≥40 in subjects with negative results at pre-vaccination (HI titer <10) or an increase of at least 4 times in HI titer for individuals with positive results at pre-vaccination (HI titer >10) at Day 22 and Day 43 in comparison to the pre-vaccination result.
Difference in Seroprotection Rates by Visit (Vaccine with Adjuvant - Vaccine without Adjuvant) | 13 months after vaccination (Day 22, Day 43, Day 133, Day 223, Day 403)
  The primary objective of this study is to determine the optimal influenza vaccination strategy in patients with HIV infection.
  Comparisons were made by vaccine group using differences in the percentage of subjects with seroprotection and were presented with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Centro Médico São Francisco, Curitiba, Paraná
  - ICG - Instituto Centro de Genomas, São Paulo, São Paulo

REFERENCES:
- [Background] Clark TW, Pareek M, Hoschler K, Dillon H, Nicholson KG, Groth N, Stephenson I. Trial of 2009 influenza A (H1N1) monovalent MF59-adjuvanted vaccine. N Engl J Med. 2009 Dec 17;361(25):2424-35. doi: 10.1056/NEJMoa0907650. Epub 2009 Sep 10. PMID 19745215
- [Background] Novel Swine-Origin Influenza A (H1N1) Virus Investigation Team; Dawood FS, Jain S, Finelli L, Shaw MW, Lindstrom S, Garten RJ, Gubareva LV, Xu X, Bridges CB, Uyeki TM. Emergence of a novel swine-origin influenza A (H1N1) virus in humans. N Engl J Med. 2009 Jun 18;360(25):2605-15. doi: 10.1056/NEJMoa0903810. Epub 2009 May 7. PMID 19423869
- [Background] Evison J, Farese S, Seitz M, Uehlinger DE, Furrer H, Muhlemann K. Randomized, double-blind comparative trial of subunit and virosomal influenza vaccines for immunocompromised patients. Clin Infect Dis. 2009 May 15;48(10):1402-12. doi: 10.1086/598193. PMID 19361304
- [Background] Fine AD, Bridges CB, De Guzman AM, Glover L, Zeller B, Wong SJ, Baker I, Regnery H, Fukuda K. Influenza A among patients with human immunodeficiency virus: an outbreak of infection at a residential facility in New York City. Clin Infect Dis. 2001 Jun 15;32(12):1784-91. doi: 10.1086/320747. Epub 2001 May 16. PMID 11360221
- [Background] Kunisaki KM, Janoff EN. Influenza in immunosuppressed populations: a review of infection frequency, morbidity, mortality, and vaccine responses. Lancet Infect Dis. 2009 Aug;9(8):493-504. doi: 10.1016/S1473-3099(09)70175-6. PMID 19628174
- [Background] Ranieri R, Veronelli A, Santambrogio C, Pontiroli AE. Impact of influenza vaccine on response to vaccination with pneumococcal vaccine in HIV patients. AIDS Res Hum Retroviruses. 2005 May;21(5):407-9. doi: 10.1089/aid.2005.21.407. PMID 15929703
- [Background] Sullivan PS, Hanson DL, Dworkin MS, Jones JL, Ward JW; Adult and Adolescent Spectrum of HIV Disease Investigators. Effect of influenza vaccination on disease progression among HIV-infected persons. AIDS. 2000 Dec 1;14(17):2781-5. doi: 10.1097/00002030-200012010-00018. PMID 11125897
- [Background] Tasker SA, Treanor JJ, Paxton WB, Wallace MR. Efficacy of influenza vaccination in HIV-infected persons. A randomized, double-blind, placebo-controlled trial. Ann Intern Med. 1999 Sep 21;131(6):430-3. doi: 10.7326/0003-4819-131-6-199909210-00006. PMID 10498559
- [Background] Yamanaka H, Teruya K, Tanaka M, Kikuchi Y, Takahashi T, Kimura S, Oka S; HIV/Influenza Vaccine Study Team. Efficacy and immunologic responses to influenza vaccine in HIV-1-infected patients. J Acquir Immune Defic Syndr. 2005 Jun 1;39(2):167-73. PMID 15905732